CLINICAL TRIAL: NCT02587403
Title: A Randomized, Prospective Study Comparing Fortiva™ Porcine Dermis vs. Strattice™ Reconstructive Tissue Matrix in Patients Undergoing Complex Open Primary Ventral Hernia Repair
Brief Title: A Comparison of Fortiva and Strattice Tissue Matrices in Complex, Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTI-2015-02
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fortiva™ Porcine Dermis (Active Comparator): Fortiva Porcine Dermis implantation during repair of complex ventral hernia
  Interventions: Device: Fortiva™ Porcine Dermis
- Strattice™ Reconstructive Tissue Matrix (Active Comparator): Strattice tissue matrix implanted during repair of complex ventral hernia
  Interventions: Device: Strattice™ Reconstructive Tissue Matrix

INTERVENTIONS:
Device: Fortiva™ Porcine Dermis — Fortiva Porcine Dermis implantation during repair of complex ventral hernia
  Arms: Fortiva™ Porcine Dermis
Device: Strattice™ Reconstructive Tissue Matrix — Strattice tissue matrix implanted during repair of complex ventral hernia
  Arms: Strattice™ Reconstructive Tissue Matrix

SUMMARY:
The objective of this study is to compare the effectiveness of Fortiva Porcine Dermis versus Strattice Reconstructive Tissue Matrix for the underlay reinforcement of complex ventral hernia repair and assess post-operative complication rates, long term hernia recurrence rates.

DETAILED DESCRIPTION:
This is a randomized, prospective, double-blinded study evaluating the efficacy of Fortiva Porcine Dermis versus Strattice Reconstructive Tissue Matrix in 120 patients with large complex abdominal wall ventral hernias undergoing single stage repair. The patient will be blinded to treatment as well as an independent qualified evaluator to confirm evidence of reoccurrence. This post-market study compares two FDA cleared biologic hernia materials. Fortiva™ porcine dermis, processed by RTI Surgical, Inc., a non-cross linked porcine dermis will be compared to Strattice™ Reconstructive Tissue Matrix by Life Cell, a non-cross linked porcine dermis for reinforcement during the single stage open reconstruction of abdominal wall defects. The primary outcome will be hernia recurrence at 1 year. Outcomes will be evaluated at 6 weeks, 3 months, 6 months and 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Have a BMI < or equal to 40
* Have a pre-operative estimated hernia defect of 200 cm2 OR multiple hernia defects whose combined area is ≥ an estimated 200 cm2. Patients whose defects do NOT meet or exceed 200 cm2 intra-operatively will be withdrawn from the study and will be considered an intra-operative screen failure
* Have no contraindications to the test material (s)
* Have a life expectancy greater than 1 year in the opinion of the Investigator
* Able to provide informed consent
* Able and willing to return for scheduled study visits over 2 years post-operatively (following research related surgery)

Exclusion Criteria:

* < 18 years of age
* Subject is determined to have an American Society of Anesthesiologists'(ASA) physical class of 4, 5, or 6
* Have a BMI >40
* Have a hernia estimated to be <200 cm2
* Have abdominal loss of domain such that the operation would be impractical or would adversely affect respiratory or cardiovascular function to an unacceptable degree in the opinion of the investigator
* Inability to close the fascia primarily without abdominal wall mobilization or component separation
* Participation in an investigational drug or device study that would impact the safety or scientific integrity of this study (in the opinion of the Investigator and with the approval of the Sponsor) within the past 6 weeks prior to enrollment into this trial
* Have active necrotizing fasciitis or any other known active local or systemic infection
* Have a known collagen metabolism disorder or any medical condition that could interfere with normal tissue healing process as determined by the Investigator
* Have a known active malignancy present and/or had chemotherapy 12 weeks prior to screening or planned chemotherapy within 12 weeks of enrollment with exception of BCC or SCC
* Have known moderate to severe cirrhosis which in the opinion of the Investigator would impact the outcome of this trial
* Have a life expectancy less than 1 year
* Be unable to participate in the informed consent process
* Be unable or unwilling to return for scheduled study visits over the 2 year post-operative assessment period
* Received high dose steroids (>/=100mg of prednisone) within the past 6 weeks
* Known tobacco use within the past 6 weeks or positive serum cotinine test at time of admission
* Uncontrolled diabetes (i.e. known HbA1C value > 7% within the last 6 weeks)
* History of drug addiction (recreational drugs, prescription drugs or alcohol) that in the Investigator's opinion may interfere with protocol assessments and/or the subject's ability to complete the required follow up
* Pregnancy and/or breastfeeding
* Enterocutaneous fistula
* Ventral hernia repairs involving active infection
* Inability to obtain primary fascial closure (Intra-operatively)
* Planned use of external VAC dressing intra-operatively

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Bochicchio, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix
Started | 60 | 60
Completed | 51 | 44
Not Completed | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.5) | 59.2 (13.1) | 59.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 27 | 62
  Male | 25 | 33 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 50 | 51 | 101
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (4.7) | 32.3 (5.4) | 32 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Experience a True Hernia Recurrence
Description: True hernia recurrence as diagnosed by physical exam or CT scan
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix
Number analyzed (Participants) | 60 | 60
Participants | 2 | 1

2. Secondary Outcome: SF-36 MCS
Description: SF-36 mental component summary scale ranges from 0-100. Higher score indicates better self reported health.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix
Number analyzed (Participants) | 54 | 49
score on a scale | 48.9 (9.2) | 48.9 (9.2)

3. Secondary Outcome: Pain Measured Using the Visual Analog Scale for Pain
Description: Visual analog scale measures extremes of pain on a scale from 0-10. 0 is no pain and 10 is worst pain
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix
Number analyzed (Participants) | 54 | 49
units on a scale | 2.41 (2.22) | 2.37 (2.32)

4. Secondary Outcome: True Recurrence at 24 Months
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix
Number analyzed (Participants) | 55 | 52
Participants | 3 | 1

5. Secondary Outcome: Time to Discharge
Description: Time is from date of procedure to date of each patient discharge. Mean of each group is provided
Time Frame: Discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix
Number analyzed (Participants) | 55 | 53
Days | 7.93 (2.32) | 8.11 (3.39)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Site reported adverse events
Arm/Group | Fortiva™ Porcine Dermis | Strattice™ Reconstructive Tissue Matrix
All-Cause Mortality (participants affected / at risk) | 0/60 | 5/60
Serious Adverse Events (participants affected / at risk) | 13/60 | 23/60
Other Adverse Events (participants affected / at risk) | 25/60 | 23/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fortiva™ Porcine Dermis (N=60) | Strattice™ Reconstructive Tissue Matrix (N=60)
Seroma (Infections and infestations) | 3 | 0
Abdominal Wall Infection (Infections and infestations) | 1 | 1
Atrial fibrillation with RVR (Cardiac disorders) | 0 | 1
Abdominal Pain (General disorders) | 0 | 1
Acute Kidney Injury (Endocrine disorders) | 0 | 1
Acute Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHOLECOCHOLITHIASIS (Gastrointestinal disorders) | 0 | 1
Dehydration (General disorders) | 0 | 2
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Dizziness (General disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Endocarditis (Cardiac disorders) | 0 | 1
Fluid Collection (Injury, poisoning and procedural complications) | 0 | 1
Fluid Overload (Injury, poisoning and procedural complications) | 0 | 1
GI Bleed (Gastrointestinal disorders) | 1 | 1
Headache (General disorders) | 0 | 1
Hematoma (Injury, poisoning and procedural complications) | 0 | 1
Hyponatremia (General disorders) | 1 | 0
Intra abdominal abscess (Injury, poisoning and procedural complications) | 0 | 3
Intra abdominal fluid collection (Injury, poisoning and procedural complications) | 1 | 1
Multisystem organ failure (General disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pain (Injury, poisoning and procedural complications) | 1 | 0
Partial small bowel obstruction (Gastrointestinal disorders) | 0 | 1
PICC line infection (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Progressive Atherosclerotic (Cardiac disorders) | 0 | 1
Pulmonary embolism (General disorders) | 1 | 0
Recurrent GI bleed (Gastrointestinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Small bowel obstruction (Gastrointestinal disorders) | 2 | 4
Subcarinal mass with metastis to brain (General disorders) | 0 | 1
Symptomatic bradycardia (Cardiac disorders) | 0 | 1
Third degree AV block (Cardiac disorders) | 0 | 1
Valve infection (Cardiac disorders) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fortiva™ Porcine Dermis (N=60) | Strattice™ Reconstructive Tissue Matrix (N=60)
Abdominal cellulitis (Infections and infestations) | 1 | 4
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 2
Constipation (General disorders) | 2 | 2
Hallucinations (General disorders) | 2 | 0
Hypocalcemia (General disorders) | 2 | 0
Hyphosphatemia (General disorders) | 2 | 2
Itching (General disorders) | 0 | 2
Nausea (Injury, poisoning and procedural complications) | 3 | 2
Open wound (Injury, poisoning and procedural complications) | 3 | 0
Post op pain (Injury, poisoning and procedural complications) | 6 | 2
Seroma (General disorders) | 6 | 11
Urinary tract infection (Renal and urinary disorders) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 4 | 3
Wound infection (Injury, poisoning and procedural complications) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT02587403/Prot_SAP_000.pdf